CLINICAL TRIAL: NCT04605939
Title: Clinical Application of Fibroblast Activation Protein PET/MRI for Diagnosis and Staging in Liver Fibrosis
Brief Title: Clinical Application of Fibroblast Activation Protein PET/MRI in Liver Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoli Lan, Director of the Department of nuclear medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0507
Record Dates: First submitted 2020-10-25; First posted 2020-10-28 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Liver Fibrosis; Positron Emission Tomography; Magnetic Resonance Imaging
MeSH Terms: conditions — Liver Cirrhosis | interventions — Positron-Emission Tomography; Magnetic Resonance Spectroscopy; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTA-FAPI PET/MR (Experimental): Investigators select subjects from patients with suspected or diagnosed or treated lievr fibrosis for 68Ga-DOTA-FAPI PET/MR imaging.
  Interventions: Device: PET/MR; Device: PET/CT

INTERVENTIONS:
Device: PET/MR — Each subject undergoes PET/MR imaging within 40-60 minutes after injection.
  Other Names: Positron Emission Tomography/Magnetic Resonance
Device: PET/CT — Each subject undergoes PET/CT imaging within 40-60 minutes after injection.
  Other Names: Positron Emission Tomography/Computed Tomography

SUMMARY:
Positron Emission Tomography (PET) provides a valuable tool for the diagnosis and staging of liver fibrosis. Activation of hepatic stellate cell (HSC) is a key link in the pathophysiological development of liver fibrosis. In human liver tissue, fibroblast activation protein (FAP) was only expressed in active HSCs and fibroblasts, but not in static HSCs. Therefore, FAP has become an excellent target for diagnosis and treatment of liver fibrosis. Recently, radionuclide-labeled fibroblast activation protein inhibitors (FAPI) as a new novel positron tracer has shown to be effective to detect various cancers. In this prospective study, the investigators will use the most advanced imaging equipments, integrated PET/MR, and PET/CT with gallium-68 (68Ga) -FAPI to image patients with or suspected of liver fibrosis, the aim is to explore the value of 68Ga-FAPI hybrid PET/MR and PET/CT in liver fibrosis.

DETAILED DESCRIPTION:
Liver fibrosis is a key step in the development of various chronic liver diseases (viral hepatitis, alcoholic liver disease, non-alcoholic fatty liver disease, autoimmune liver disease, etc.) to cirrhosis and an important link that affects the prognosis of chronic liver disease. Fibrosis is histologically reversible, and early liver fibrosis can still be reversed to restore liver tissue to normal. However, due to the lack of specific initial symptoms and accurate non-invasive diagnostic methods, the onset of liver fibrosis is insidious. Most patients have developed liver cirrhosis and/or hepatocellular carcinoma when they are diagnosed, and some even require liver transplantation. If liver fibrosis can be diagnosed accurately and treated early, the prognosis of chronic liver disease can be improved.

Positron Emission Tomography (PET) provides a valuable tool for the diagnosis and staging of liver fibrosis. Activation of hepatic stellate cell (HSC) is a key link in the pathophysiological development of liver fibrosis. In human liver tissue, fibroblast activation protein (FAP) was only expressed in active HSCs and fibroblasts, but not in static HSCs. Therefore, FAP has become an excellent target for diagnosis and treatment of liver fibrosis. Recently, radionuclide-labeled fibroblast activation protein inhibitors (FAPI) as a new novel positron tracer has shown to be effective to detect various cancers. In this prospective study, the investigators will use the most advanced imaging equipments, integrated PET/MR, and PET/CT with gallium-68 (68Ga) -FAPI to image patients with or suspected of liver fibrosis, the aim is to explore the value of 68Ga-FAPI hybrid PET/MR and PET/CT in liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or diagnosed or treated liver fibrosis.
* Subjects are able to understand and sign the informed consent voluntarily, with good compliance.

Exclusion Criteria:

* Acute systemic diseases and electrolyte disorders.
* Pregnant or lactating women.
* Patients refuse to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 68Ga-DOTA-FAPI PET/MR for diagnosis and staging in liver fibrosis. | 2 years
  For 100 subjects with suspected or diagnosed or treated liver fibrosis who have completed 18F-FDG PET/CT imaging, diagnosis and staging results of 68Ga-DOTA-FAPI PET/MR, PET/CT will be compared to transient elastography（TE）, pathology, clinical and follow-up result.
Correlation of 68Ga-DOTA-FAPI PET/MR parameters and liver fibrosis progression. | 2 years
  Analyze the correlation between the parameters displayed by 68Ga-DOTA-FAPI PET/MR and the pathological staging of liver fibrosis, serological scores, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China

REFERENCES:
- [Derived] Song Y, Qin C, Chen Y, Ruan W, Gai Y, Song W, Gao Y, Hu W, Qiao P, Song X, Lv X, Zheng D, Chu H, Jiang D, Yang L, Lan X. Non-invasive visualization of liver fibrosis with [68Ga]Ga-DOTA-FAPI-04 PET from preclinical insights to clinical translation. Eur J Nucl Med Mol Imaging. 2024 Oct;51(12):3572-3584. doi: 10.1007/s00259-024-06773-z. Epub 2024 Jun 8. PMID 38850311
- [Derived] Qin C, Song Y, Liu X, Gai Y, Liu Q, Ruan W, Liu F, Hu F, Lan X. Increased uptake of 68Ga-DOTA-FAPI-04 in bones and joints: metastases and beyond. Eur J Nucl Med Mol Imaging. 2022 Jan;49(2):709-720. doi: 10.1007/s00259-021-05472-3. Epub 2021 Jul 9. PMID 34241652
- [Derived] Zhang X, Song W, Qin C, Liu F, Lan X. Non-malignant findings of focal 68Ga-FAPI-04 uptake in pancreas. Eur J Nucl Med Mol Imaging. 2021 Jul;48(8):2635-2641. doi: 10.1007/s00259-021-05194-6. Epub 2021 Jan 15. PMID 33452634